CLINICAL TRIAL: NCT03183245
Title: A Phase 3 Study to Compare the Efficacy and Safety of Humacyte's Human Acellular Vessel With That of an Autologous Arteriovenous Fistula in Subjects With End Stage Renal Disease
Brief Title: Comparison of the Human Acellular Vessel (HAV) With Fistulas as Conduits for Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Humacyte, Inc. (Industry)
Collaborators: CTI Clinical Trial and Consulting Services (Other); California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLN-PRO-V007
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2024-11

CONDITIONS: Renal Failure; End Stage Renal Disease; Hemodialysis; Vascular Access
MeSH Terms: conditions — Renal Insufficiency; Kidney Failure, Chronic | interventions — Arteriovenous Shunt, Surgical; Renal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Human Acellular Vessel (HAV) (Experimental): The HAV is a tissue-engineered vascular conduit (6mm diameter) for hemodialysis access in patients with end-stage renal disease. It will be surgically implanted in the forearm or upper arm on Study Day 0.
  Interventions: Biological: Human Acellular Vessel (HAV); Other: Hemodialysis
- Arteriovenous fistula (AVF) (Active Comparator): The comparator is an autologous arteriovenous fistula created in the forearm or upper arm on Study Day 0.
  Interventions: Procedure: Arteriovenous fistula (AVF); Other: Hemodialysis

INTERVENTIONS:
Biological: Human Acellular Vessel (HAV) — Surgical implantation of the HAV and subsequent use of the implanted vascular conduit for hemodialysis vascular access.
  Arms: Human Acellular Vessel (HAV)
Procedure: Arteriovenous fistula (AVF) — Surgical creation of an autologous arteriovenous fistula and subsequent use of the implanted vascular conduit for hemodialysis vascular access.
  Arms: Arteriovenous fistula (AVF)
Other: Hemodialysis — Procedure that filters a person's blood when their kidneys are no longer functioning properly

SUMMARY:
The main purpose of this study is to compare the Human Acellular Vessel (HAV) with arteriovenous fistula (AVF) when used for hemodialysis access

DETAILED DESCRIPTION:
This is a Phase 3, prospective, multicenter, open-label, randomized, two-arm, comparative study. Subjects who sign informed consent will undergo study-specific screening assessments within 45 days from the day of informed consent.

Eligible study subjects will be randomized to receive either an HAV or AVF. The randomization will be stratified by upper arm or forearm placement based on the investigator's determination of where the study access (SA) should be located. Subjects will be followed to 24 months post SA creation at routine study visits regardless of patency status. After 24 months, AVF subjects with a patent SA will be followed (while the SA remains patent) for up to 5 years (60 months) post SA creation at routine study visits. After 24 months, HAV subjects will be followed (regardless of SA patency) for 5 years (60 months) post SA creation at routine study visits.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with end-stage renal disease (ESRD), receiving HD via DC and are suitable for the creation of an AVF or implantation of AVG for HD access.
2. Subjects who plan to undergo HD at a dialysis unit of a participating dialysis provider for at least the first 6 months after SA creation.
3. Subjects aged at least 18 years at Screening.
4. Suitable anatomy for creation of a forearm or upper arm AVF and for implantation of straight or looped HAV in either the forearm or upper arm.
5. Hemoglobin ≥8 g/dL and platelet count ≥100,000 /mm3.
6. International Normalized Ratio (INR) ≤ 1.5.
7. Female subjects must be either:

   1. Of non-childbearing potential, which is defined as post-menopausal (at least 1 year without menses prior to Screening) or documented surgically sterile or post hysterectomy (at least 1 month prior to Screening).
   2. Or, of childbearing potential, in which case:

   i. Must have a negative urine or serum pregnancy test at Screening, and ii. Must agree to use at least one form of the following birth control methods for the duration of the study:
   * Established use of oral, injectable or implanted hormonal methods of contraception.
   * Placement of an intrauterine device or intrauterine system.
   * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/ gel/ film/ cream/ suppository.
8. Subject, or legal representative, able to communicate effectively with investigative staff, competent and willing to give written informed consent, and able to comply with entire study procedures including all scheduled follow-up visits.
9. Life expectancy of at least 2 years.

Exclusion Criteria:

1. Subjects who are optimal candidates for radiocephalic AVF as indicated by meeting ALL of the following criteria:

   1. No previous failed AVF.
   2. Cephalic vein diameter on ultrasound of more than 3.5mm.
   3. Radial artery diameter on ultrasound of more than 3mm.
   4. Vein depth of less than 0.5cm from the skin.
   5. Normal Allen's test indicating that ulnar artery flow to the hand is sufficient.
   6. No calcification in the wall of the distal radial artery.
   7. Sufficient length of the proposed fistula outflow vein to provide an adequate (at least 6 cm) cannulation segment.
   8. No evidence of iatrogenic injury to target artery or vein.
2. Uncontrolled diabetes;

   a. HbA1c >10% (at Screening).
3. History or evidence of severe peripheral arterial disease in the extremity selected for implant.
4. Known or suspected central vein stenosis or obstruction on the side of planned SA creation, unless corrected prior to randomization.
5. Planned AVF creation that requires more than one stage to complete. (e.g. basilic vein transposition AVF performed in 2 stages).
6. Planned AVF creation by means other than suture or vascular anastomotic clips (e.g. endovascular surgery or other anastomotic creation devices).
7. Treatment with any investigational drug or device within 60 days prior to study entry (Day 0) or ongoing participation in a clinical trial of an investigational product.
8. Cancer that is actively being treated with a cytotoxic agent.
9. Documented hyper-coagulable state.
10. Bleeding diathesis.
11. Active clinically significant immune-mediated disease, not controlled by maintenance immunosuppression.

    1. Low dose glucocorticoid therapy (e.g. 5-10mg prednisone [Deltason]) is acceptable.
    2. High dose glucocorticoid therapy for treatment of autoimmune flare, or other inflammatory diseases is excluded.
    3. Patients using glucocorticoids for immunosuppression post-transplant to prevent against transplanted allograft rejection in the period post allograft failure are excluded.
    4. The following examples of immunosuppressive agents (or the like) are exclusionary for enrollment in this clinical trial:

       * tacrolimus or FK506 [Prograf]
       * mycophenolate mofetil [Cellcept],
       * cyclosporine [Sandimmune or Gengraf]
       * sirolimus [Rapamune] (this only includes systemically administered, drug eluting stents are acceptable)
12. Anticipated renal transplant within 6 months.
13. History of heparin-induced thrombocytopenia.
14. Venous outflow from SA cannot be located more centrally than the venous outflow of any previous failed access in that extremity.
15. Active local or systemic infection (white blood cells [WBC] > 15,000 cells/mm3 at Screening). If the infection resolves, the subject must be at least one week post resolution of that infection before SA creation.
16. Known serious allergy or intolerance to aspirin and alternative antiplatelet therapy.
17. Pregnant women, or women intending to become pregnant during the course of the trial.
18. Any other condition which in the judgment of the investigator would preclude adequate evaluation of the safety and efficacy of the SA.
19. Previous enrollment in this study or any other study with HAV.
20. Employees of Humacyte and employees or relatives of an investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with functional patency at 6 months post study access (SA) creation | 6 months post SA creation
  Co-primary endpoint #1: Proportion of subjects with functional patency at 6 months post study access (SA) creation
  The definition of "functional patency" is: Dialysis with "2 needles for ≥75% of dialysis sessions over a continuous 4-week period and either: (1) 4 consecutive sessions during the 4-week period in which 2 needles are used and the mean dialysis machine blood pump speed is ≥300 mL/min, or (2) a measured spKt/Vurea is ≥ 1.4 or urea reduction ratio >70% during any session in which 2 needles are used within the 4-week period. SpKt/Vurea is calculated from pre and post-treatment serum urea nitrogen concentrations, body weight, and dialysis session duration."
  The functional patency ascertainment period will take place between the 1st day of Week 21 (Day 140) and the last day of Week 26 (Day 181) after AVF creation or HAV placement. The endpoint is met when the functional patency criteria are satisfied within any consecutive 4 week period within this ascertainment period.
Proportion of subjects with secondary patency of SA at 12 months post SA creation. | 12 months post SA creation
  Co-primary endpoint #2: Proportion of subjects with secondary patency of SA at 12 months post SA creation.
  The SA maintains secondary patency until it is abandoned, irrespective of interventions to maintain or restore patency.
  Abandonment is defined as AVF or HAV that can no longer be used for 2-needle, prescribed dialysis as it may be unable to provide adequate flows and/or is deemed unsafe for the subject, and the associated problem cannot be corrected by any intervention, including medical, surgical, or radiological interventions or rest.

SECONDARY OUTCOMES:
Time to loss of secondary patency (abandonment). | 12, 24, and 60 months post SA creation
Incidence rate of HD access related interventions over the period from SA creation until SA abandonment or 12 months post SA creation | 12 months post SA creation
Incidence rate of infections related to any HD access in situ over the period from SA creation until 12 months post SA creation, irrespective of SA abandonment. | 12 months post SA creation
Proportion of subjects with unassisted functional patency at 6 months post SA creation. | 6 months post SA creation
Incidence rate of HD access-related interventions over the period from SA creation until SA abandonment or the conclusion of the suitability ascertainment period (6 months). | 6 months post SA creation
Time to loss of primary unassisted patency | 12, 24, and 60 months post SA creation
Proportion of HD sessions completed via DC (1 or 2 lines) over the period from SA creation until 12 months post SA creation, irrespective of SA abandonment. | 12 months post SA creation
Number of days with DC in situ "catheter contact time" over the period from SA creation until 12 months post SA creation, irrespective of SA abandonment | 12 months post SA creation
Histopathological remodeling of HAV and AVF - based on histological examination of SA samples explanted for clinical reasons | 12, 24, and 60 months post SA creation
Incidence rate of HD access-related infections over the period from SA creation until SA abandonment. | 12, 24, and 60 months post SA creation
Incidence rate of clinically significant aneurysm or pseudoaneurysm over the period from SA creation until SA abandonment | 12, 24, and 60 months post SA creation
Incidence rate of SA site infections (CDC definition) over the period from SA creation until SA abandonment. | 12, 24, and 60 months post SA creation
Frequency and severity of AEs. | 12, 24, and 60 months post SA creation

CONTACTS AND LOCATIONS:
Overall Officials: Shamik Parikh, MD, Study Director — Humacyte, Inc.
Locations (31):
- United States (31):
  - Arizona Kidney Disease and Hypertension Center (AKDHC), Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - University of California, Irvine, Irvine, California
  - University of California San Diego, Jacobs Medical Center, La Jolla, California
  - University of CA, San Diego - LaJolla VA Hospital, La Jolla, California
  - Alliance Research, Laguna Hills, California
  - VA Long Beach Healthcare System, Long Beach, California
  - University of Southern California, Los Angeles, California
  - Huntington Hospital, Pasadena, California
  - UC Davis, Sacramento, California
  - Balboa Nephrology, San Diego, California
  - Mills Peninsula Hospital, San Mateo, California
  - Olive View- UCLA Medical Center, Sylmar, California
  - Denver Health Medical Center, Denver, Colorado
  - The Vascular Experts, Darien, Connecticut
  - Memorial Healthcare System, Pembroke Pines, Florida
  - Coastal Vascular & Interventional, PLLC, Pensacola, Florida
  - Tampa General Hospital, Tampa, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Decatur Memorial Hospital, Decatur, Illinois
  - United Surgical Associates, Lexington, Kentucky
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Kidney Care & Transplant Services of New England, West Springfield, Massachusetts
  - Rutgers University, Newark, New Jersey
  - Overlook Medical Center, Summit, New Jersey
  - Surgical Specialists of Charlotte, Charlotte, North Carolina
  - Kaiser Permanente Sunnsyide, Portland, Oregon
  - VA Pittsburgh, Pittsburgh, Pennsylvania
  - The Regional Medical Center, Orangeburg, South Carolina
  - University of Tennessee Knoxville, Knoxville, Tennessee
  - South Plains Surgery Center, Lubbock, Texas

IPD SHARING:
Plan to Share IPD: No